CLINICAL TRIAL: NCT06204822
Title: Non-contact Blood Pressure and SpO2 Measurement Based on Image Sensor
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202301108RINC
Record Dates: First submitted 2024-01-03; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Blood Pressure; SpO2

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- blood pressure measurement: 1. Participants sit in a comfortable posture with hands naturally placed on the table or thighs, palms facing up without obstruction, facing the camera lens. Rest for 2 minutes.
  2. First blood pressure measurement is taken, and images and data are recorded for 2 minutes.
  3. Participants place both feet on a stool, exerting pressure on the instep (hooking towards the knee) for 1 minute.
  4. Maintain the instep pressure and perform the second blood pressure measurement, recording images and data for 2 minutes.
  5. Participants place both feet flat on the ground, resting for 1 minute.
  6. Third blood pressure measurement is taken, and images and data are recorded for 2 minutes.
  7. The examiner adjusts the program settings, and the participant repeats steps 2 to 6 once.
- blood oxygen saturation measurement: 1. Participants sit in a comfortable posture with both hands placed naturally on the table or thighs, palms facing up without obstruction, and facing the camera lens. They rest for 2 minutes.
  2. Participants breathe normally while recording images and data for 1 minute.
  3. Participants hold their breath until discomfort (aiming for at least 40 seconds) while recording images and data for 1 minute.
  4. Participants return to normal breathing, and images and data are recorded for 3 minutes.
  5. The experimenter adjusts program settings, and participants repeat steps 2 to 4 once.

SUMMARY:
This study aims to develop an automated and real-time non-contact vital sign measurement system using cameras. It will collaborate with physicians from National Taiwan University Hospital to conduct measurements during outpatient visits or hospitalizations. This allows physicians to non-invasively measure multiple vital signs (such as heart rate, blood pressure, and oxygen saturation) upon your entry to the outpatient clinic or hospital. Simultaneously, the measurements will be verified using commercially available contact-based instruments. The research outcomes of this project aim to enhance the convenience, safety, and comfort of vital sign measurements for outpatient visits, hospitalizations, and long-term care in the future.

DETAILED DESCRIPTION:
The experiment of this project is to use a camera to measure blood pressure, blood oxygen saturation and pulse, record images of the face and hands, and use the image processing algorithm we developed to extract the signals from the images to estimate blood pressure and blood oxygen Concentration and pulse values. The experimental process will be carried out in accordance with the "experimental setup, blood pressure measurement, and blood oxygen saturation measurement" process. At the same time, commercially available measurement instruments will be used to conduct clinical experiments and verification. The experimental setup diagram is shown in Figure 1. Blood pressure and blood pressure The oxygen saturation measurement process is shown in Figure 2. The blood pressure measurement process takes about 10 minutes, and the blood oxygen measurement process takes about 5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-85 years old
* Install the physiological measurement device on people who do not feel any physical discomfort

Exclusion Criteria:

* Age > 85 years, age < 18 years
* Patients with arrhythmia
* Those with a history of severe heart disease
* Those who wear makeup on their face (for example: foundation cream, sunscreen lotion, foundation...etc.).
* The body will make involuntary, short-term, rapid or repetitive movements unconsciously, resulting in the inability to control the body to reach a stable and static state. For example: patients with motor-related Tourette Syndrome, etc.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 200 subjects from National Taiwan University Hospital and National Taiwan University of Science and Technology are expected to be included.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-03-06 (Estimated); Study Completion 2026-03-06 (Estimated)

PRIMARY OUTCOMES:
Blood pressure changes | 10 min
  Use OMRON HEM-7157T to record changes in blood pressure values
Blood oxygen changes | 5 min
  Use Cntec CMS-50E to record changes in blood pressure values

CONTACTS AND LOCATIONS:
Overall Officials: Huang TZU-JU, M.S., Principal Investigator — NTUST
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided